CLINICAL TRIAL: NCT06411470
Title: Gastrointestinal Microflora and Serum Metabolomics in Patients With Pancreatic Cancer and Chronic Pancreatitis
Status: Recruiting | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Xiangyu Kong, Principle Investigator, Changhai Hospital
Other Study IDs: CHEC2024-149
Record Dates: First submitted 2024-05-01; First posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Pancreatic Cancer; Chronic Pancreatitis
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatitis, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- pancreatic cancer: Pathologic diagnosis of pancreatic ductal adenocarcinoma
- chronic pancreatitis: Diagnosis of CP defined as having obvious morphological features of CP (i.e., the presence of pancreatic calcifications on CT scan and/or magnetic resonance cholangiopancreatography)
- healthy people: Other benign disease populations without pancreatic lesions

SUMMARY:
The investigators plan to collect throat swabs, saliva, feces and serum samples from pancreatic cancer patients, chronic pancreatitis patients and healthy people and clarify the characteristics of oral flora and serum metabolome of pancreatic cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1.Pathologic diagnosis of pancreatic ductal adenocarcinoma；Diagnosis of CP defined as having obvious morphological features of CP (i.e., the presence of pancreatic calcifications on CT scan and/or magnetic resonance cholangiopancreatography)；Other benign disease populations without pancreatic lesions.

Exclusion Criteria:

1. Pregnant women.
2. Patients with coagulation disorders who are unable to undergo blood tests.
3. Have a history of using antibiotics or probiotics within the past 3 months.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: pancreatic cancer,chronic pancreatitis,healthy people
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-04-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
serum metabolites | Baseline
  Perform Untargeted liquid chromatography-tandem mass spectrometry (LC-MS/MS) to analyse serum samples collected from pancreatic cancer patients, chronic pancreatitis patients and healthy people.
Gastrointestinal microbiota | Baseline
  Perform 16S RNA sequence and shotgun metagenomic analysis of fecal, throat swabs and salivary samples collected from pancreatic cancer patients, chronic pancreatitis patients and healthy people.
Overall Survival | up to 2 years
  The length of time (in days) from study enrollment that participants remain alive.
Predictive model | up to 2 years
  Combined with preoperative imaging and pathological information, a predictive model of pancreatic cancer would be established based on the metabolic and microbiota difference. Verify the stability and accuracy of our model in larger cohorts and promote clinical translation.

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China